CLINICAL TRIAL: NCT02209740
Title: A Prospective, Cohort Study of Renal and Bone Outcome After Changing Tenofovir in Patients With Renal Toxicity According to Antiretroviral Strategy
Brief Title: Renal and Bone Outcome After Switching Tenofovir to Different Antiretroviral Strategies
Acronym: TDFOUT
Status: Completed | Type: Observational
Sponsor: Asociacion para el Estudio de las Enfermedades Infecciosas (Network)
Responsible Party: Principal Investigator, Jose L. Casado, Clinical Investigator, Asociacion para el Estudio de las Enfermedades Infecciosas
Other Study IDs: TDFOUT; 218/12 revised (Other: CEIC)
Record Dates: First submitted 2014-08-02; First posted 2014-08-06 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Renal Disease
Keywords: renal toxicity, HIV, antiretroviral, outcome
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tenofovir switch: Patients switched tenofovir to different antiretroviral regimen according to physicians decision
  Interventions: Other: Tenofovir switch

INTERVENTIONS:
Other: Tenofovir switch — Patients switched tenofovir to different antiretroviral regimen according to physicians decision

SUMMARY:
Renal outcome could be different after switching tenofovir to different antiretroviral strategies, in case of renal toxicity. Therefore, it is necessary to evaluate the importance of renal evolution in these patients, in terms of grade and time to renal improvement, according to the different options after interrupting tenofovir. The aim of this study was to explore the renal outcome after tenofovir according to new antiretroviral regimen.

DETAILED DESCRIPTION:
Renal toxicity has become an important issue in a large number of HIV infected patients receiving a tenofovir-containing regimen. However, there are no data about the best antiretroviral regimen in patients switching tenofovir because of renal toxicity, in time, grade or persistence of renal improvement. Thus, patients with renal toxicity on tenofovir, defined as:

* a progressive decrease of at least 25% of estimated glomerular filtration rate (GFR, by chronic kidney disease-epi equation), or
* confirmed value of GFR below 60 ml/min in two successive determinations, or
* proximal tubular renal dysfunction, as indicated by the presence of at least 3 of the following parameters: proteinuria> 150 mg/g; excretion fractional of phosphorus in urine > 20%; glucosuria > 150 mg; or/and tubular proteinuria/albuminuria ratio above 0.4.

who changed to the combination of abacavir plus a third drug, or to a nucleoside analogues-free antiretroviral combination (dual therapy, monotherapy) will be followed for 1 year to establish the time and grade of improvement (defined as the lack of above criteria).

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients
* Older than 18 years
* Receiving a Tenofovir-containing regimen, and with criteria of renal toxicity (see above)
* Switching the antiretroviral regimen

Exclusion Criteria:

* Pregnancy
* Patients receiving prolonged therapy with other nephrotoxic drugs
* Patients not receiving or interrupting antiretroviral regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients in regular clinical and analytical follow up, receiving a tenofovir-containing regimen
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Renal outcome | 48 weeks
  Evolution of renal parameters after switching tenofovir according to antiretroviral drug or regimen used, in terms of GFR (glomerular filtration rate by Chronic Kidney Disease-epidemiological collaboration equation) improvement, increase in excretion fractional of phosphorus in urine, decrease in proteinuria, and in glycosuria. As control group, renal outcome will be evaluated in patients continuing TDF-based therapy

SECONDARY OUTCOMES:
Antiviral efficacy | 48 weeks
  Number of patients without virological failure, defined as an HIV RNA level above 37 copies/ml, 48 weeks after the change of tenofovir
Bone mineral density (BMD) changes | 48 weeks
  Changes in BMD in the subgroup of patients with two successive BMD measurements, before and after TDF switch, according to baseline risk factors for BMD change (age, body mass index, hypovitaminosis D, secondary hyperparathyroidism), in comparison with patients continuing TDF

OTHER OUTCOMES:
Antiviral safety | 48 weeks
  Number (and percentage) and degree of adverse events, and percentage of therapy withdrawal, according to antiretroviral strategy after the change of tenofovir

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Casado, MD, Principal Investigator — Asociacion para el Estudio de las Enfermedades Infecciosas
Locations (1):
- Hospital Ramon y Cajal, Madrid, Spain